CLINICAL TRIAL: NCT02523391
Title: A Phase I, Randomised, Open-label Cross-over Bioequivalence Study of Capsule and Tablet Formulations of TA-8995 in Healthy Male Subjects
Brief Title: Bioequivalence Study of Capsule and Tablet Formulations of TA-8995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TA-8995-08
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Dyslipidaemia
MeSH Terms: conditions — Dyslipidemias | interventions — TA-8995

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Period 1 (Experimental): Either 5mg TA-8995 Capsule or Tablet
  Interventions: Drug: TA-8995
- Treatment Period 2 (Experimental): Either 5mg TA-8995 Capsule or Tablet
  Interventions: Drug: TA-8995

INTERVENTIONS:
Drug: TA-8995 — Capsule
Drug: TA-8995 — Tablet

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of capsule and tablet formulations of TA-8995 in healthy male subjects aged 18 to 55 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-55
* Body Mass Index (BMI) between 18.0 and 32.0 kg/m2, inclusive

Exclusion Criteria:

* Subject has a known hypersensitivity to any of the inactive ingredients of the study treatments.
* Subject has any other condition which, in the Investigator's opinion will interfere with the study.
* Subjects who are still participating in another clinical study (eg, attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) within 3 months or 5 half-lives (whichever is longer) prior to the first dose in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of TA-8995 capsule and tablet formulations | 72 hours
Peak Plasma Concentration (Cmax) of TA-8995 capsule and tablet formulations | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom